CLINICAL TRIAL: NCT06676566
Title: Information, Follow-up and Early Diagnosis of Children at Risk for Type 1 Diabetes
Acronym: iT1D
Status: Enrolling by invitation | Type: Observational
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: iT1D/2024
Record Dates: First submitted 2024-10-28; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Type 1 Diabetes Mellitus; Stage 2 Type 1 Diabetes; Stage 1 Type 1 Diabetes; Stage 3 Type 1 Diabetes
Keywords: type 1 diabetes; genetic risk; islet autoantibodies; staging of type 1 diabetes; islet autoimmunity; children; follow-up; autoantibody screening
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Genetic risk without islet autoantibodies: This group has more than 10% risk of early onset of islet autoimmunity and can come to visits at 2, 6 and 10 years of age. At the visits blood samples are drawn and disease risk information and information about symptoms is given. The child will wear an accelerometer for one week after each visit.
- Genetic risk with 1 islet autoantibody: This group will be followed annually up to diabetes diagnosis or to 18 years of age. At the visits blood samples are drawn and disease risk information and information about symptoms is given. The child will wear an accelerometer for one week after each visit.
- Genetic risk with multiple islet autoantibodies: This group will come to visits every three months up to diagnosis or 18 years of age. At the visits blood samples are drawn and disease risk information and information about symptoms is given. An OGTT will be performed at some of the visits. The child will wear an accelerometer and a CGM for one week after each visit.
- Children with stage 3 type 1 diabetes who have taken part in the study before diagnosis: Annual visits at the study center will continue for the first 5 years after diagnosis.

SUMMARY:
The aim is to investigate whether screening for islet autoantibodies, regular follow-up, and increased knowledge in families about the progression of the disease in children at high genetic risk or with single or multiple islet autoantibodies (stage 1 or 2 type 1 diabetes) ensures an earlier diagnosis of stage 3 type 1 diabetes compared to no screening or follow-up.

Risk factors studied in relation to disease progression are the impact of higher-than-average weight gain, insulin resistance, and physical activity, both individually and in combination, on the risk of developing autoantibodies and disease progression.

An alternative diagnostic method, continuous glucose monitoring (CGM), will be evaluated for its for usefullness in early diagnosis of stage 2 and 3 type 1 diabetes as alternatives to oral glucose tolerance tests.

Another aim is to investigate the psychological impact of being aware that the children are at a higher risk of type 1 diabetes.

When a child in the study develops stage 3 type 1 diabetes, the psychological impact and metabolic control during the first five years after diagnosis will be compared to children not followed before the diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Children 0 -10 years with high or moderate genetic risk of type 1 diabetes, measured by a combined analysis of HLA and non-HLA SNPs. Moderate genetic risk is defined as 8-10% risk of developing multiple islet autoantibodies before 6 years of age, and high genetic risk as over 10% risk of developing multiple islet autoantibodies before 6 years of age.
* Children 0-18 years of age screened in other research studies or tested at a clinical site and found to have a single autoantibody (before stage 1 type 1 diabetes) or multiple islet autoantibodies without or with impaired glucose tolerance (stage 1 or 2 type 1 diabetes, respectively).
* Children will be invited to participate in the current study if they have moderate or high genetic risk and 1) have participated in a prevention trial but have dropped out or the trial has ended 2) are not willing to participate in prevention trial.
* Children screened and found to be positive for islet autoantibodies in other studies (TEDDY, TrialNet, Innodia etc) or in clinical settings but which have not progressed to stage 3 type 1 diabetes can also be invited to participate in the current study.

Exclusion Criteria:

* Stage 3 type 1 diabetes
* Currently participating in a prevention study

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who have been screened for genetic risk for type 1 diabetes at birth in the ASTR1D study and other children who have been screened for either genetic risk or islet autoantibodies in other studies.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2034-10-01 (Estimated); Study Completion 2034-10-01 (Estimated)

PRIMARY OUTCOMES:
Early diabetes diagnosis, measured as HbA1c, symptoms, incidence of DKA | From enrollment to a maximum of 10 years follow-up
  Investigate if screening for islet autoantibodies, regular follow-up and increased knowledge in the families regarding progression of the disease in children at high genetic risk or with single or multiple islet autoantibodies (stage 1 or 2 type 1 diabetes) ensures an early diagnosis of stage 3 type 1 diabetes, measured by HbA1c and symptoms, and prevents DKA as compared to no screening or follow-up.
  The hypothesis is that screening and follow-up ensures an early diagnosis with no/few symptoms and prevents DKA.
Growth in relation to development of 1 islet autoantibody and progression to multiple islet autoantibodies and clinical type 1 diabetes | From enrollement to a maximum of 10 years follow up.
  Investigate the impact of higher-than-average weight gain (SDS body weight in kg) on the risk of developing islet autoantibodies, progressing from one to several autoantibodies (stage 1 or 2 type 1 diabetes) and to progression to clinical type 1 diabetes (stage 3 type 1 diabetes). The hypothesis is that higher than average weight gain increase the risk of islet autoimmunity.
Insulin resistance in relation to development of islet autoantibodies, progression to multiple islet autoantibodies and clinical type 1 diabetes | From enrollment to a maximum of 10 years follow-up
  Investigate the impact insulin resistance, measured as HOMA-IR on the risk of developing islet autoantibodies, progression from a single islet autoantibody to multiple islet autoantibodies (stage 1 or 2 type 1 diabetes) and to stage 3 clinical type 1 diabetes. The hypothesis is that higher insulin resistance, measured as HOMA-IR, increase the risk of developing islet autoantibodies and the rate of progression to multiple islet autoantibodies and stage 3 type 1 diabetes.
Physical activity in relation to development of islet autoantibodies, progression to multiple islet autoantibodies and clinical type 1 diabetes | From enrollement to a maximum of 10 years follow up.
  Investigate the impact of physical activity, measured by summary statistics from an accelerometer worn during 1 week/year on the risk of developing islet autoantibodies and progress to multiple islet autoantibodies and clinical type 1 diabetes. The hypothesis is that increased time and intensity of physical activity decreases the risk of islet autoimmunity and the rate of progression to multiple islet autoantibodies and type 1 diabetes.
Measurements derived from continous glucose monitoring (CGM) compared to blood glucose testing during OGTT in diagnosing early stages of type 1 diabetes | From enrollment to a maximum of 10 years follow-up
  Investigate different methods of an early diagnosis of stage 2 and 3 type 1 diabetes as alternative options for oral glucose tolerance tests. Measurements derived from continuous glucose monitoring (CGM), such as mean glucose, standard deviation, interquartile range, coefficient of variation, Time in Range (TIR), Time Below Range (TBR), Low Blood Glucose Index (LBGI), Mean Amplitude of Glycemic Excursions (MAGE) will be used. The hypothesis is that CGM data can be interpreted and summarized using one or more summary statistics for which specific cut-off values could be defined and validated, which could be used in the clinic replacing the need for performing OGTT.
Psychological impact of screening and follow up, measured by validated questionnaires | From enrollment to a maximum of 10 years follow-up
  Investigate the psychological impact of being aware that the child is at a higher risk of type 1 diabetes, as measured by anxiety levels, study satisfaction, compliance with screening and follow-up, with respect to having first degree relatives with type 1 diabetes, demographic and socioeconomic factors. The hypothesis is that factors associated with anxiety can be identified, and that anxiety and satisfaction can be improved by providing parents with adequate information, especially in parents more prone to developing anxiety
Psychological impact of screening after diagnosis measured by validated questionnaires | From T1D diagnosis until the last visit, maximum 5 years after diagnosis.
  Investigate the psychological impact during the first 5 years after a diagnosis of stage 3 type 1 diabetes in children previously followed in the study compared to children not followed before the diagnosis. The hypothesis is that screening and follow-up and an early diagnosis of type 1 diabetes improves coping in the families.
Metabolic control after clinical diagnosis | From T1D diagnosis until the last visit, maximum 5 years after diagnosis.
  Investigate the metabolic control (measured by HbA1c (mmol/mol), fasting and stimulated C-peptide and data derived from CGM (mean glucose, SD)) during the first 5 years after a diagnosis of stage 3 type 1 diabetes in children previously followed in the study compared to children not followed before the diagnosis. The hypothesis is that screening and follow-up and an early diagnosis of type 1 diabetes improves metabolic control during at least the first 5 years after diagnosis. For the metabolic control, the national diabetes registry data will be used as a reference group.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Elding Larsson, MD, PhD, Prof., Principal Investigator — Lund University
Locations (1):
- CRC Jan Waldenströms gata 35, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Number of particiants and if they have genetic risk, single or multiple autoantibodies (stage 2 type 1 diabetes) and number diagnosed with stage 3 type 1 diabetes